CLINICAL TRIAL: NCT00048074
Title: A Randomized, Double-blind Study Comparing the Effect of Different Treatment Regimens of Intravenous Bonviva on Lumbar Bone Mineral Density in Women With Osteoporosis
Brief Title: DIVA Study - A Study of Different Regimens of Intravenous Administration of Bonviva (Ibandronate) in Women With Post-Menopausal Osteoporosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BM16550
Record Dates: First submitted 2002-10-24; First posted 2002-10-25 (Estimated); Results first posted 2016-02-03 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: Post Menopausal Osteoporosis
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Ibandronic Acid

ARMS (3):
- 1 (Experimental): oral placebo daily and IV ibandronate 2 mg q 2 mo
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 2 (Experimental): oral ibandronate 2.5 mg daily and IV placebo q 2 mo and q 3 mo
  Interventions: Drug: ibandronate [Bonviva/Boniva]
- 3 (Experimental): oral placebo daily and IV ibandronate 3 mg q 3 mo
  Interventions: Drug: ibandronate [Bonviva/Boniva]

INTERVENTIONS:
Drug: ibandronate [Bonviva/Boniva] — 2mg iv every 2 months
  Arms: 1
Drug: ibandronate [Bonviva/Boniva] — 2.5mg po daily
  Arms: 2
Drug: ibandronate [Bonviva/Boniva] — 3mg iv every 3 months
  Arms: 3

SUMMARY:
This study will assess the efficacy and safety of intravenous administration of Bonviva regimens in women with post-menopausal osteoporosis, compared to oral daily administration. Patients will also receive daily supplementation with vitamin D and calcium. The anticipated time of study treatment is 2+ years, and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* women 55-80 years of age;
* post-menopausal for >=5 years;
* ambulatory.

Exclusion Criteria:

* malignant disease diagnosed within the previous 10 years (except basal cell cancer that has been successfully removed);
* breast cancer within the previous 20 years;
* allergy to bisphosphonates;
* previous treatment with an intravenous bisphosphonate at any time;
* previous treatment with an oral bisphosphonate within the last 6 months, >1 month of treatment within the last year, or >3 months of treatment within the last 2 years.

Ages: 55 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1395 (Actual)
Dates: Start 2002-06; Primary Completion 2005-05 (Actual); Study Completion 2005-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (62):
- United States (19):
  - Little Rock, Arkansas
  - Irvine, California
  - Rancho Mirage, California
  - Leesburg, Florida
  - Gainesville, Georgia
  - Coeur d'Alene, Idaho
  - Bethesda, Maryland
  - St Louis, Missouri
  - Billings, Montana
  - Omaha, Nebraska
  - Albuquerque, New Mexico
  - New York, New York
  - Bismarck, North Dakota
  - Fargo, North Dakota
  - Wyomissing, Pennsylvania
  - Rapid City, South Dakota
  - San Antonio, Texas
  - Virginia Beach, Virginia
  - Madison, Wisconsin
- Australia (5):
  - Darlinghurst
  - Melbourne
  - Nedlands
  - St Leonards
  - Sydney
- Belgium (2):
  - Brussels
  - Liège
- Canada (4):
  - Toronto, Ontario
  - Laval, Quebec
  - Montreal, Quebec
  - Saskatoon, Saskatchewan
- Czechia (2):
  - Pilsen
  - Prague
- Denmark (5):
  - Aalborg
  - Aarhus
  - Ballerup Municipality
  - Copenhagen
  - Vejle
- France (2):
  - Lyon
  - Orléans
- Germany (3):
  - Berlin
  - Bochum
  - Hamburg
- Budapest, Hungary
- Italy (3):
  - Arenzano
  - Siena
  - Valeggio sul Mincio
- Mexico (2):
  - Mexico City
  - Monterrey
- Norway (3):
  - Haugesund
  - Oslo
  - Stavanger
- Poland (2):
  - Grudziądz
  - Krakow
- South Africa (3):
  - Cape Town
  - Pretoria
  - Sommerset West
- Spain (3):
  - Barcelona
  - Madrid
  - Santander
- United Kingdom (3):
  - Aberdeen
  - Manchester
  - Newcastle upon Tyne

REFERENCES:
- [Derived] Bianchi G, Czerwinski E, Kenwright A, Burdeska A, Recker RR, Felsenberg D. Long-term administration of quarterly IV ibandronate is effective and well tolerated in postmenopausal osteoporosis: 5-year data from the DIVA study long-term extension. Osteoporos Int. 2012 Jun;23(6):1769-78. doi: 10.1007/s00198-011-1793-9. PMID 21975558

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1804 participants were screened for the study, from which 1395 participants were enrolled and randomized into treatment with ibandronate. The trial was conducted at 58 centers in 16 countries from June 2002 to May 2005.
Pre-assignment Details: Out of the 1395 participants who were randomized into the study, only 1382 participants received at least one dose of trial treatment and had at least one follow-up assessment as 4 participants did not have safety follow-up and 9 participants did not receive trial treatment.
Groups:
- Ibandronate 2.5mg Daily: Participants received 2.5 milligrams (mg) of ibandronate orally daily and IV placebo injection at intervals of either 2 or 3 months for a total treatment period of 24 months.
- Ibandronate 2mg q 2 mo IV: Participants received 2 mg of ibandronate intravenously (IV) every two months and placebo tablet daily for a total treatment period of 24 months.
- Ibandronate 3mg q 3 mo IV: Participants received 3 mg of ibandronate IV every three months and placebo tablet daily for a total treatment period of 24 months.
Period: Overall Study
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Started | 465 | 448 | 469
Completed | 384 | 361 | 372
Not Completed | 81 | 87 | 97
Not completed — Adverse Event | 46 | 41 | 53
Not completed — Death | 3 | 3 | 2
Not completed — Lost to Follow-up | 2 | 6 | 6
Not completed — Withdrawal by Subject | 28 | 30 | 35
Not completed — Protocol Violation | 1 | 3 | 0
Not completed — Study participation was terminated | 0 | 1 | 0
Not completed — Husband ill | 0 | 1 | 0
Not completed — Poor compliance | 0 | 1 | 0
Not completed — Out of station | 0 | 1 | 1
Not completed — Social reasons | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population: All participants who were randomized and had at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point were included.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV | Total
Number analyzed (Participants) | 465 | 448 | 469 | 1382
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.7 (6.08) | 66.6 (6.26) | 65.8 (6.30) | 66.0 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 465 | 448 | 469 | 1382
  Male | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Relative Percent Change From Baseline in Mean Bone Mineral Density (BMD) of Lumbar Spine (L2-L4) at 12 Months
Description: BMD was measured by a single dual-energy x-ray absorptiometry (DXA) scan of the lumbar spine at the time of screening and at Month 12. The change in BMD was defined as the relative difference between the last individual measurement available at 12 months and Baseline, using the following formula: Relative change = 100 x (BMD at 1 year - BMD at Baseline) / (BMD at Baseline)
Time Frame: Baseline and Month 12
Population: Per protocol population: Participants who were randomized, received at least one dose of study medication and had at least one efficacy (BMD or serum CTX) follow-up data point and did not have any major violations of the protocol.
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 368 | 350 | 359
Percent Change | 3.8199 (3.8576) | 5.0872 (3.8746) | 4.8188 (3.7613)
Statistical Analysis 1: Comparison: Ibandronate 2.5mg Daily vs Ibandronate 2mg q 2 mo IV; The primary hypothesis was that the difference in the effects of daily oral ibandronate and IV ibandronate (2mg q 2 mo IV) on the relative change in lumbar spine BMD (L2 - L4) was small, no more than 1%, the margin of clinical equivalence; Test type: Non-Inferiority or Equivalence — The IV dosing regimen (2mg q 2 mo IV) was considered non-inferior to the 2.5 mg daily regimen if the lower bound of the two-sided 95% CI on the difference in mean percent change in BMD was greater or equal to -1 percentage point; p < 0.001, ANOVA; Mean Difference (Final Values) = 1.257, 95% CI 2-sided [0.701 to 1.814] — Treatment effect is the difference in the mean values of the IV regimen (2mg q 2 mo IV) and the active-control
Statistical Analysis 2: Comparison: Ibandronate 2.5mg Daily vs Ibandronate 3mg q 3 mo IV; The primary hypothesis was that the difference in the effects of daily oral ibandronate and IV ibandronate (3mg q 3 mo IV) on the relative change in lumbar spine BMD (L2 - L4) was small, no more than 1%, the margin of clinical equivalence; Test type: Non-Inferiority or Equivalence — The IV dosing regimen (3mg q 3 mo IV) was considered non-inferior to the 2.5 mg daily regimen if the lower bound of the two-sided 95% CI on the difference in mean percent change in BMD was greater or equal to -1 percentage point; p < 0.001, ANOVA; Mean Difference (Final Values) = 1.025, 95% CI 2-sided [0.471 to 1.578] — Treatment effect is the difference in the mean values of the IV regimen (3mg q 3 mo IV) and the active-control

2. Secondary Outcome: Relative Percent Change From Baseline in Mean BMD of Lumbar Spine (L2-L4) at 24 Months
Description: BMD was measured by a single dual-energy x-ray absorptiometry (DXA) scan of the lumbar spine at the time of screening and at Month 24. The change in BMD was defined as the relative difference between the last individual measurement available at 24 months and Baseline, using the following formula: Relative change = 100 x (BMD at 1 year - BMD at Baseline) / (BMD at Baseline)
Time Frame: Baseline and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 334 | 320 | 334
Percent Change | 4.8412 (4.8654) | 6.3999 (4.7392) | 6.2777 (5.0049)

3. Secondary Outcome: Absolute Change From Baseline in Mean BMD of Lumbar Spine (L2 - L4) at Month 12 and Month 24
Description: BMD was measured by a single dual-energy x-ray absorptiometry (DXA) scan of the lumbar spine at screening, Month 12 and Month 24. The absolute change from Baseline in mean BMD of the lumbar spine (L2-L4) was defined as the difference between the last individual measurement available at Month 12 or Month 24 and Baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Absolute Change (g/cm^2)
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Absolute Change (g/cm^2)
  Month 12, n= 368, 350, 359 | 0.028 (0.0287) | 0.037 (0.0282) | 0.035 (0.0269)
  Month 24, n= 334, 320, 334 | 0.036 (0.0361) | 0.047 (0.0347) | 0.046 (0.0357)

4. Secondary Outcome: Relative Percent Change From Baseline in BMD of Proximal Femur (Consisting of Total Hip, Trochanter, and Femoral Neck) at Month 12 and 24
Description: BMD was measured by a single DXA scan of the proximal femur at the time of screening, Month 12 and Month 24.The change in BMD of the proximal femur (total hip, trochanter, femoral neck) was defined as the relative difference between the last individual measurement available at Month 12 or Month 24and Baseline, using the following formula: Relative change = 100 x (BMD at 1 year/2year - BMD at Baseline) / (BMD at Baseline). BMD of fractured bones that could impact the scan area were not taken into account. Only participants with data available at particular timepoint were analyzed.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percent Change
  Total hip, Month 12, n = 364, 343, 357 | 1.7857 (2.8171) | 2.5150 (2.6737) | 2.3604 (3.5156)
  Total hip , Month 24, n = 330, 316, 333 | 2.2011 (3.6997) | 3.3699 (2.9749) | 3.1279 (4.5422)
  Trochanter, Month 12, n = 364, 343, 357 | 2.9721 (4.1651) | 4.0275 (3.8890) | 3.8144 (6.0921)
  Trochanter, Month 24, n = 330, 316, 333 | 3.4669 (4.7241) | 5.0428 (4.4640) | 4.9165 (7.5057)
  Femoral neck, Month 12, n = 364, 343, 357 | 1.6129 (4.1050) | 1.9700 (3.5537) | 2.3055 (3.9283)
  Femoral neck, Month 24, n = 330, 316, 333 | 2.2457 (4.3015) | 2.7449 (4.1996) | 2.7849 (4.6723)

5. Secondary Outcome: Absolute Change From Baseline in BMD of Proximal Femur (Consisting of Total Hip, Trochanter, and Femoral Neck) at Month 12 and 24
Description: BMD was measured by a single DXA scan of the proximal femur at the time of screening, Month 12 and Month 24. The absolute change in BMD was defined as the difference between the last individual measurement available at Month 12 or Month 24 and Baseline. BMD of fractured bones that could impact the scan area were not taken into account. Only participants with data available at particular timepoint were analyzed.
Time Frame: Baseline, Month 12 and Month 24
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Absolute Change (g/cm^2)
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Absolute Change (g/cm^2)
  Total hip, Month 12, n = 364, 343, 357 | 0.013 (0.0202) | 0.018 (0.0192) | 0.016 (0.0213)
  Total hip, Month 24, n = 330, 316, 333 | 0.015 (0.0259) | 0.025 (0.0211) | 0.022 (0.0278)
  Trochanter, Month 12, n = 364, 343, 357 | 0.016 (0.0229) | 0.022 (0.0209) | 0.020 (0.0250)
  Trochanter, Month 24, n = 330, 316, 333 | 0.019 (0.0256) | 0.029 (0.0242) | 0.026 (0.0322)
  Femoral neck , Month 12, n = 364, 343, 357 | 0.010 (0.0243) | 0.013 (0.0227) | 0.014 (0.0240)
  Femoral neck , Month 24, n = 330, 316, 333 | 0.014 (0.0258) | 0.018 (0.0279) | 0.018 (0.0278)

6. Secondary Outcome: Relative Change From Baseline in Serum C-telopeptide of Alpha-chain of Type I Collagen (CTX) at Month 6, 12, and 24
Description: Serum CTX, a biochemical marker of bone resorption, was measured using the Elecsys s-CTX-I assay, an electrochemiluminescence immunoassay (ECLIA) technique. Samples for serum CTX measurements were collected from participants immediately prior to their IV dosing. Thus, the values reported here represent trough or residual values taken at the end of the 2 month or 3 month IV dosing interval. The change in serum CTX was defined as the relative difference between the last individual measurement available at Month 6 or Month 12 or Month 24 and Baseline, using the following formula: Relative change = 100 x (CTX at Month 6/Month 12/Month 24- CTX at Baseline) / (CTX at Baseline). Only participants with data available at particular timepoint were analyzed.
Time Frame: Baseline, At Month 6, 12, and 24.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percent Change
  Month 6, n = 358, 342, 345 | -54.715 (30.2820) | -55.539 (42.6206) | -51.196 (31.0579)
  Month 12, n = 360, 342, 347 | -54.387 (33.2810) | -48.042 (95.3711) | -49.873 (36.0415)
  Month 24, n = 310, 301, 298 | -51.549 (35.0888) | -41.338 (76.8201) | -44.325 (38.1338)

7. Secondary Outcome: Absolute Change From Baseline in Serum CTX at Month 6, 12, and 24
Description: Serum CTX, a biochemical marker of bone resorption, was measured using the Elecsys s-CTX-I assay, an electrochemiluminescence immunoassay (ECLIA) technique. Samples for serum CTX measurements were collected from participants immediately prior to their IV dosing. Thus, the values reported here represent trough or residual values taken at the end of the 2 month or 3 month IV dosing interval. The absolute change from Baseline in serum CTX was defined as the difference between the last individual measurement available at Month 6 or Month 12 or Month 24 and Baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: Baseline, At Month 6, 12, and 24.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Absolute Change (ng/mL)
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Absolute Change (ng/mL)
  Month 6, n = 358, 342, 345 | -0.318 (0.2550) | -0.322 (0.2015) | -0.281 (0.2018)
  Month 12, n = 360, 342, 347 | -0.321 (0.2624) | -0.318 (0.2239) | -0.290 (0.2196)
  Month 24, n = 310, 301, 298 | -0.324 (0.2693) | -0.285 (0.2092) | -0.276 (0.2323)

8. Secondary Outcome: Percentage of Participants With Mean Lumbar Spine (L2 - L4) BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean lumber spine (L2 - L4) BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 368, 350, 359 | 85.1 | 92.3 | 91.6
  Above baseline, Month 24, n = 334, 320, 334 | 84.7 | 92.8 | 92.8

9. Secondary Outcome: Percentage of Participants With Total Hip BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean total hip BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 364, 343, 357 | 74.5 | 86.0 | 82.6
  Above baseline, Month 24, n = 330, 316, 333 | 77.0 | 88.6 | 85.6

10. Secondary Outcome: Percentage of Participants With Trochanter BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean trochanter BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 364, 343, 357 | 76.6 | 88.6 | 86.3
  Above baseline, Month 24, n = 330, 316, 333 | 80.0 | 92.1 | 88.6

11. Secondary Outcome: Percentage of Participants With Femoral Neck BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean femoral neck BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 364, 343, 357 | 65.1 | 74.1 | 70.0
  Above baseline, Month 24, n = 330, 316, 333 | 67.6 | 77.5 | 76.6

12. Secondary Outcome: Percentage of Participants With Mean Total Hip and Lumbar Spine BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean total hip and mean lumbar spine BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 363, 343, 355 | 66.9 | 80.5 | 76.3
  Above baseline, Month 24, n = 330, 314, 332 | 68.8 | 83.1 | 80.1

13. Secondary Outcome: Percentage of Participants With Mean Trochanter and Lumbar Spine BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean trochanter and lumbar spine BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 363, 343, 355 | 68.0 | 83.4 | 79.7
  Above baseline, Month 24, n = 330, 314, 332 | 70.9 | 85.7 | 83.1

14. Secondary Outcome: Percentage of Participants With Mean Femoral Neck and Lumbar Spine BMD Above or Equal to Baseline at Month 12 and 24
Description: A participant is a responder if the mean femoral neck and lumbar spine BMD had remained the same or increased above baseline. Only participants with data available at particular timepoint were analyzed.
Time Frame: At Month 12 and 24
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 375 | 350 | 364
Percentage of participants
  Above baseline, Month 12, n = 363, 343, 355 | 58.4 | 69.4 | 64.5
  Above baseline, Month 24, n = 330, 314, 332 | 59.7 | 72.3 | 71.7

15. Secondary Outcome: Number of Participants Who Experienced Any Adverse Events (AEs) or Serious Adverse Events (SAEs)
Description: An AE is any untoward medical occurrence in a participant or clinical investigation subject administered a pharmaceutical product and which does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE is any untoward medical occurrence that at any dose results in death, are life threatening, requires hospitalization or prolongation of hospitalization or results in disability/incapacity, and congenital anomaly/birth defect.
Time Frame: Approximately 2 years
Population: Safety Population: All participants who were randomized and had at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point.
Measure: Number; unit: participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 465 | 448 | 469
participants
  Any AE | 408 | 397 | 400
  Any SAE | 67 | 73 | 62

16. Secondary Outcome: Number of Participants With Any Marked Abnormality in Laboratory Parameters
Description: Marked laboratory test value abnormalities (high and low) are those which exceed the marked reference range (i.e., a reference range greater than the standard reference range) and which also represents a clinically relevant change from baseline of at least a designated amount. The indicated abnormal laboratory parameters (along with their marked reference range) are as follows: low and high Hematocrit (0.36 - 0.60 fraction), low and high hemoglobin (11.0 - 20.0 g/dL), low and high platelets (100 - 700 * 10^9/L), low and high white blood cell (WBC) (3.0 - 18.0 * 10^9/L), high alanine aminotransferase (ALAT) (0 - 60 U/L), high blood urea nitrogen (BUN) (0 - 14.3 mmol/L) , high creatinine (0 - 154 mmol/L), low albumin (27.0 - 48.0 g/L), low and high chloride (95 - 115 mmol/L), low potassium (3.0 - 6.0 mmol/L), low sodium (130 - 150 mmol/L), high calcium (2.00 - 2.90 mmol/L), low and high phosphate (0.75 - 1.60 mmol/L).
Time Frame: Approximately 2 years
Population: Safety Population: All participants who were randomized and had at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point. Only participants with data available for the indicated laboratory abnormality were analyzed.
Measure: Number; unit: participants
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Number analyzed (Participants) | 465 | 448 | 469
participants
  Hematocrit - High, n = 453, 433, 456 | 0 | 0 | 1
  Hematocrit - low, n = 453, 433, 456 | 0 | 2 | 5
  Hemoglobin - High, n = 453, 433, 456 | 0 | 1 | 1
  Hemoglobin - Low n = 453, 433, 456 | 2 | 5 | 5
  Platelets - High, n = 452, 431, 455 | 0 | 2 | 1
  Platelets - Low, n = 452, 431, 455 | 2 | 0 | 1
  WBC - High, n = 453, 433, 456 | 0 | 1 | 2
  WBC - Low, n = 453, 433, 456 | 4 | 4 | 2
  ALAT (SGPT) - High, n = 453, 434, 456 | 13 | 12 | 18
  BUN - High, n = 453, 434, 456 | 1 | 2 | 0
  Creatinine - High, n = 453, 434, 456 | 0 | 2 | 0
  Albumin - Low, n = 453, 434, 456 | 0 | 1 | 0
  Chloride - High, n = 453, 433, 456 | 1 | 0 | 0
  Chloride - Low, n = 453, 433, 456 | 4 | 3 | 3
  Potassium - Low, n = 453, 433, 456 | 0 | 1 | 0
  Sodium - Low, n = 453, 433, 456 | 0 | 1 | 1
  Calcium - High, n = 453, 434, 456 | 0 | 1 | 0
  Phosphate - High, n = 453, 434, 456 | 7 | 4 | 6
  Phosphate - Low, n = 453, 434, 456 | 6 | 3 | 2

ADVERSE EVENTS:
Time Frame: Approximately 2 years
Description: SAEs and non-serious AEs were reported for members of the safety population, comprised of participants who were randomized and had at least one dose of study drug, whether withdrawn prematurely or not, and who had at least one follow-up data point.
Arm/Group | Ibandronate 2.5mg Daily | Ibandronate 2mg q 2 mo IV | Ibandronate 3mg q 3 mo IV
Serious Adverse Events (participants affected / at risk) | 67/465 | 73/448 | 62/469
Other Adverse Events (participants affected / at risk) | 301/465 | 316/448 | 284/469
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 2.5mg Daily (N=465) | Ibandronate 2mg q 2 mo IV (N=448) | Ibandronate 3mg q 3 mo IV (N=469)
Abscess limb (Infections and infestations) | 0 | 1 | 0
Bronchopneumonia (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Furuncle (Infections and infestations) | 0 | 1 | 0
Klebsiella bacteraemia (Infections and infestations) | 0 | 1 | 0
Periorbital cellulitis (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0
Postoperative infection (Infections and infestations) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1
Tuberculosis (Infections and infestations) | 0 | 0 | 1
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 2 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Benign neoplasm of thyroid gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Gallbladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Myelofibrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Neuroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Non-hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Oesophageal squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Ovarian adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Ovarian cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Small cell lung cancer stage unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 2 | 3 | 1
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 0 | 0 | 2
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1
Wrist fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Drug toxicity (Injury, poisoning and procedural complications) | 1 | 0 | 0
Extradural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Meniscus lesion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Muscle injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pelvic fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Postoperative constipation (Injury, poisoning and procedural complications) | 0 | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 0 | 0 | 1
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vascular graft occlusion (Injury, poisoning and procedural complications) | 0 | 0 | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1 | 0 | 0
Gastric ulcer (Gastrointestinal disorders) | 0 | 2 | 1
Gastritis (Gastrointestinal disorders) | 1 | 0 | 2
Colonic stenosis (Gastrointestinal disorders) | 0 | 2 | 0
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 0
Rectocele (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0
Diverticulum (Gastrointestinal disorders) | 1 | 0 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0
Oesophageal ulcer (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1
Subileus (Gastrointestinal disorders) | 0 | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 4 | 2
Angina pectoris (Cardiac disorders) | 1 | 1 | 2
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 2
Arrhythmia (Cardiac disorders) | 0 | 1 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 2 | 0
Cardiac failure (Cardiac disorders) | 0 | 1 | 1
Myocardial ischaemia (Cardiac disorders) | 1 | 1 | 0
Angina unstable (Cardiac disorders) | 1 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Cardiovascular disorder (Cardiac disorders) | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1 | 0
Mitral valve disease (Cardiac disorders) | 0 | 1 | 0
Sick sinus syndrome (Cardiac disorders) | 1 | 0 | 0
Tricuspid valve incompetence (Cardiac disorders) | 0 | 1 | 0
Ventricular arrhythmia (Cardiac disorders) | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 1 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1 | 2
Cerebral infarction (Nervous system disorders) | 0 | 0 | 2
Sciatica (Nervous system disorders) | 0 | 1 | 1
Syncope (Nervous system disorders) | 1 | 0 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0 | 0
Cerebral circulatory failure (Nervous system disorders) | 0 | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0 | 0
Cerebrovascular insufficiency (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0
Epilepsy (Nervous system disorders) | 0 | 1 | 0
Grand mal convulsion (Nervous system disorders) | 0 | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1 | 0
Migraine (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 0 | 0 | 1
Reversible ischaemic neurological deficit (Nervous system disorders) | 0 | 1 | 0
Spinal vascular disorder (Nervous system disorders) | 0 | 0 | 1
Temporal lobe epilepsy (Nervous system disorders) | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal polyps (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 3 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0
Bunion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Dupuytren's contracture (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Polymyalgia rheumatica (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 1 | 1
Bile duct stone (Hepatobiliary disorders) | 2 | 0 | 1
Cholecystitis chronic (Hepatobiliary disorders) | 2 | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Ovarian cyst (Reproductive system and breast disorders) | 3 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 2 | 0
Vaginal prolapse (Reproductive system and breast disorders) | 0 | 1 | 1
Fallopian tube cyst (Reproductive system and breast disorders) | 0 | 1 | 0
Vaginal pain (Reproductive system and breast disorders) | 0 | 0 | 1
Cataract (Eye disorders) | 0 | 1 | 2
Iridocyclitis (Eye disorders) | 2 | 0 | 0
Hypotony of eye (Eye disorders) | 0 | 0 | 1
Open angle glaucoma (Eye disorders) | 1 | 0 | 0
Retinal artery thrombosis (Eye disorders) | 1 | 0 | 0
Retinal degeneration (Eye disorders) | 0 | 0 | 1
Arterial occlusive disease (Vascular disorders) | 1 | 0 | 0
Arteriosclerosis (Vascular disorders) | 0 | 1 | 0
Femoral artery occlusion (Vascular disorders) | 0 | 0 | 1
Hypertensive crisis (Vascular disorders) | 0 | 0 | 1
Hypotension (Vascular disorders) | 0 | 0 | 1
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Temporal arteritis (Vascular disorders) | 1 | 0 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1
Venous insufficiency (Vascular disorders) | 1 | 0 | 0
Cystocele (Renal and urinary disorders) | 0 | 1 | 0
Diabetic nephropathy (Renal and urinary disorders) | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0
Stress incontinence (Renal and urinary disorders) | 0 | 1 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 1 | 0
Goitre (Endocrine disorders) | 0 | 1 | 0
Hyperparathyroidism primary (Endocrine disorders) | 1 | 0 | 0
Toxic nodular goitre (Endocrine disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 0 | 1 | 0
International normalised ratio increased (Investigations) | 0 | 1 | 0
Red blood cell sedimentation rate increased (Investigations) | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 0
Diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 1
Diabetes mellitus non-insulin-dependent (Metabolism and nutrition disorders) | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 1 | 0
Histrionic personality disorder (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 1 | 0
Drug hypersensitivity (Immune system disorders) | 1 | 0 | 0
Sarcoidosis (Immune system disorders) | 1 | 0 | 0
Angioneurotic oedema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Vestibular neuronitis (Ear and labyrinth disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ibandronate 2.5mg Daily (N=465) | Ibandronate 2mg q 2 mo IV (N=448) | Ibandronate 3mg q 3 mo IV (N=469)
Nasopharyngitis (Infections and infestations) | 65 | 66 | 43
Influenza (Infections and infestations) | 51 | 43 | 35
Bronchitis (Infections and infestations) | 23 | 28 | 22
Urinary tract infection (Infections and infestations) | 28 | 24 | 18
Gastroenteritis (Infections and infestations) | 24 | 19 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 56 | 62 | 58
Arthralgia (Musculoskeletal and connective tissue disorders) | 50 | 55 | 56
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 19 | 26 | 30
Pain in extremity (Musculoskeletal and connective tissue disorders) | 16 | 27 | 18
Bone pain (Musculoskeletal and connective tissue disorders) | 8 | 23 | 11
Abdominal pain upper (Gastrointestinal disorders) | 33 | 24 | 29
Dyspepsia (Gastrointestinal disorders) | 28 | 28 | 23
Constipation (Gastrointestinal disorders) | 27 | 33 | 18
Diarrhoea (Gastrointestinal disorders) | 18 | 23 | 20
Nausea (Gastrointestinal disorders) | 25 | 22 | 13
Hypertension (Vascular disorders) | 54 | 44 | 47
Hypercholesterolaemia (Metabolism and nutrition disorders) | 32 | 29 | 19
Headache (Nervous system disorders) | 21 | 27 | 21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights